CLINICAL TRIAL: NCT02462109
Title: Catatonia in Ugandan Children With Nodding Syndrome and Effects of Treatment With Lorazepam: A Pilot Study
Brief Title: Catatonia in Nodding Syndrome and Lorazepam Treatment
Acronym: CINS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HS 1330
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Catatonia; Nodding Syndrome
MeSH Terms: conditions — Catatonia; Nodding Syndrome | interventions — Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lorazepam (Experimental): Children with confirmed Nodding syndrome that had 2 or more of the symptoms on the 10-item Kampala Catatonia Panel (KCP) scale were recruited to undergo the catatonia test using oral Lorazepam EG® (n.v. Eurogenerics s.a. Brussels, Belgium) using the 1 mg formulation tablets. The amount of Lorazepam (LZP) drug given orally was based on the weight of the child. The lower dose (0.5 mg) was used as starting dose for patients with <30 kg body weight, while the higher dose (1 mg) as the starting dose for patients with >30 kg body weight.
  A positive response to a catatonia test consisted of a reduction in catatonic symptoms, 60 minutes later, by at least 50% assessed by the KCP (using all 10 items). If no response to the initial dose of LZP, was observed after one hour, a second administration of the same medication at double the dose was given. Catatonia was again assessed at 60 minutes thereafter. If no response was observed, the test was considered negative.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — Lorazepam was given based on the weight of the child with Catatonia. The lower dose (0.5 mg) was used as starting dose for patients with <30 kg body weight, while the higher dose (1 mg) as the starting dose for patients with >30 kg body weight.
  Other Names: Ativan

SUMMARY:
Nodding Syndrome is an enigmatic neuropsychiatric syndrome affecting children and adolescents mostly in Eastern Africa. The symptoms of Nodding Syndrome and catatonia seem to overlap. The researchers' objectives in this study were to investigate the presence and types of catatonic symptoms in children with Nodding Syndrome and observe their response to one or two doses of lorazepam, the first-line treatment for catatonia.

DETAILED DESCRIPTION:
In this pilot study, the investigators examined a convenient sample of children and adolescents with Nodding Syndrome (NS) for catatonic symptoms using standardized criteria. The investigators also tested whether oral lorazepam (LZP) administered to those who qualified to have pediatric catatonia would alleviate symptoms. This was a cross-sectional descriptive study of catatonia in NS patients in Northern Uganda and an exploratory study of using one or two doses of lorazepam as a catatonia test.

All the children with confirmed NS that had 2 or more of symptoms of catatonia were recruited to undergo the catatonia test using oral Lorazepam EG® (n.v. Eurogenerics s.a. Brussels, Belgium) using the 1 mg formulation tablets. It was proposed to perform a catatonia test using Lorazepam (LZP) as first choice medication, as this is the medication that has been used most commonly in pediatric catatonia.

The amount of drug given was based on the weight of the child. The lower dose (0.5 mg) was used as starting dose for patients with <30 kg body weight, while the higher dose (1 mg) as the starting dose for patients with >30 kg body weight.

A positive response to a catatonia test consisted of a reduction in catatonic symptoms, 30 or 60 minutes later, by at least 50% .Positive responses were documented by video footage before and after administration of LZP.

If no response to the initial dose of LZP, was observed after one hour, a second administration of the same medication at double the dose was given. Catatonia was again assessed at 30 and 60 minutes thereafter. If no response was observed, the test was considered negative.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents with Nodding Syndrome as defined by the consensus definition agreed upon in the international Nodding Syndrome research meeting held in Kampala, Uganda July 2012.
2. Presence of two or more catatonic items on the Kampala Catatonia Panel.
3. Written informed consent from caregiver.

Exclusion Criteria:

1. Children and adolescents with Nodding Syndrome who had a history of having used a benzodiazepine drug in the past 48 hours prior to intervention.
2. Children and adolescents with Nodding Syndrome who had a concurrent acute illness (e.g febrile illness, pneumonia) at time of assessment.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
A positive catatonia test (>50% reduction in catatonia symptoms and signs) on the responses of the children and adolescents with Nodding Syndrome and catatonia to test doses of oral Lorazepam. | Measured at 60 minutes after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Kakooza-Mwesige, MMed, Principal Investigator — Makerere University College of Health Sciences, Kampala, Uganda; Dirk M Dhossche, MD, PhD, Study Director — University of Mississippi Medical Center, Jackson, USA

REFERENCES:
- [Background] Smith SL, Grelotti DJ, Fils-Aime R, Uwimana E, Ndikubwimana JS, Therosme T, Severe J, Dushimiyimana D, Uwamariya C, Bienvenu R, Alcindor Y, Eustache E, Raviola GJ, Fricchione GL. Catatonia in resource-limited settings: a case series and treatment protocol. Gen Hosp Psychiatry. 2015 Jan-Feb;37(1):89-93. doi: 10.1016/j.genhosppsych.2014.10.009. Epub 2014 Oct 30. PMID 25467078
- [Background] Tibrewal P, Narayanaswamy J, Zutshi A, Srinivasaraju R, Math SB. Response rate of lorazepam in catatonia: a developing country's perspective. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Dec 1;34(8):1520-2. doi: 10.1016/j.pnpbp.2010.08.017. Epub 2010 Sep 8. PMID 20804808
- [Background] Kakooza-Mwesige A, Wachtel LE, Dhossche DM. Catatonia in autism: implications across the life span. Eur Child Adolesc Psychiatry. 2008 Sep;17(6):327-35. doi: 10.1007/s00787-008-0676-x. Epub 2008 Apr 21. PMID 18427869
- [Background] Sejvar JJ, Kakooza AM, Foltz JL, Makumbi I, Atai-Omoruto AD, Malimbo M, Ndyomugyenyi R, Alexander LN, Abang B, Downing RG, Ehrenberg A, Guilliams K, Helmers S, Melstrom P, Olara D, Perlman S, Ratto J, Trevathan E, Winkler AS, Dowell SF, Lwamafa D. Clinical, neurological, and electrophysiological features of nodding syndrome in Kitgum, Uganda: an observational case series. Lancet Neurol. 2013 Feb;12(2):166-74. doi: 10.1016/S1474-4422(12)70321-6. Epub 2013 Jan 8. PMID 23305742
- [Background] Dhossche DM. Decalogue of catatonia in autism spectrum disorders. Front Psychiatry. 2014 Nov 6;5:157. doi: 10.3389/fpsyt.2014.00157. eCollection 2014. No abstract available. PMID 25414675
- [Derived] Kakooza-Mwesige A, Dhossche DM, Idro R, Akena D, Nalugya J, Opar BT. Catatonia in Ugandan children with nodding syndrome and effects of treatment with lorazepam: a pilot study. BMC Res Notes. 2015 Dec 28;8:825. doi: 10.1186/s13104-015-1805-5. PMID 26710961